CLINICAL TRIAL: NCT05847959
Title: The Relationship Between XinKang-I and Chronic Heart Failure: Protocol for a Randomized Controlled Study.
Brief Title: The Relationship Between XinKang-I and Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dongguan Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jianfeng Ye, Head of Cardiology, Dongguan Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DongguanHTCM
Record Dates: First submitted 2023-04-13; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Traditional Chinese Medicine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): The intervention group will receive not only Western medicine, but also XK-I. The therapeutic drugs used in the control group will be according to the European Society of Cardiology's 2021 guidelines for the diagnosis and treatment of acute and chronic heart failure.
  Interventions: Drug: Traditional Chinese medicine prescription：XinKang-I
- The control group (No Intervention): The control group will receive Western medicine.The therapeutic drugs used in the control group will be according to the European Society of Cardiology's 2021 guidelines for the diagnosis and treatment of acute and chronic heart failure.

INTERVENTIONS:
Drug: Traditional Chinese medicine prescription：XinKang-I — XK-I will be used in intervention group (20 grams of radix astragalus, 20 grams of radix codonopsis, 10 grams of stir-fried semen lepidii, 8 grams of sweet apricot kernel, 10 grams of cassia twig, 15 grams of poria cocos, 10 grams of atractylodes, 5 grams of honey-roasted licorice, 15 grams of radix et rhizoma salviae miltiorrhizae, 10 grams of chuanxiong rhizoma, 5 grams of tangerine peel).Patients will take XK-I once a day, divided into morning and evening administration. The treatment lasted for 8 weeks.
  Arms: intervention group

SUMMARY:
Background: Heart failure is the severe and terminal stage of various heart diseases, which is characterized by high morbidity, mortality and readmission. There are few studies on the relationship between XinKang-I(XK-I) and chronic heart failure.

Objective: To explore the relationship between XK-I and chronic heart failure. Methods/design: The trial is a single-center, single-blind, randomized study (1:1). It will recruit 110 patients with chronic heart failure who syndrome of qi deficiency yang deficiency and blood stasis. The intervention group will receive not only Western medicine, but also XK-I. The primary end points will be the changes in oxygen consumption volume of anaerobic threshold (VO2AT), maximum oxygen volume uptake (VO2max), and 6-minute walking distance after 8 weeks of treatment. Both groups will receive 8 weeks of treatment.

Ethics and dissemination: Ethical approval was granted by Ethics Committee of Dongguan TCM Hospital. Results will be disseminated via peer-reviewed publications and presentations at international conferences.

ELIGIBILITY:
Inclusion Criteria:

1. History of CHF or clinical findings of CHF for more than 3 months. CHF was diagnosed in accordance with the European Society of Cardiology's 2021 Guidelines for the Diagnosis and Treatment of Acute and Chronic Heart Failure.
2. Patients ranged in age from 18 to 85.
3. Cardiac function was graded at grade II-IV (New York Heart Association functional class).
4. Patients who had not used traditional Chinese medicine for treating heart failure within 1 week before enrollment;
5. Written informed consent will be obtained.

Exclusion Criteria:

1. acute cardiac insufficiency, acute myocarditis, severe valvular heart disease, malignant arrhythmia, obstructive cardiomyopathy, pericardial tamponade, constrictive pericarditis or acute coronary syndrome
2. severe lung, liver or kidney dysfunction
3. nervous and hematopoietic system
4. malignant tumors
5. hemodynamic nstability
6. pulmonary embolism
7. severe infection
8. pregnant or lactating
9. refusal to provide written informed consent for this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes in 6-minute walking distance(distance, meter). | 8 weeks
  Cardiac function
oxygen consumption volume of anaerobic threshold (VO2AT, ml) | 8 weeks
  Cardiac function
maximum oxygen volume uptake (VO2max, ml/min) in cardiopulmonary function test | 8 weeks
  Cardiac function